CLINICAL TRIAL: NCT01421238
Title: Framing and Perinatal Decision Making at Extremes of Prematurity
Brief Title: Framing and Decision Making in Neonatology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Elke U. Weber, Jerome A. Chazen Professor of International Business and Professor of Psychology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AAAB8193
Record Dates: First submitted 2011-08-08; First posted 2011-08-22 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Prematurity; Framing; Perinatal Decision Making
Keywords: Decision Making; Premature infant; Informed consent; Prematurity; Framing; Negotiation Model
MeSH Terms: conditions — Premature Birth | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resuscitation Default Arm (Experimental): After receiving a description of an impending delivery of a 23 week gestational infant, participants in this arm were presented with the following information:
  The doctor goes on to say that at this hospital infants born at 23 weeks will receive resuscitation, unless their parents object. If you decline resuscitation please check the box below:
  Please check if you decline resuscitation []
  Interventions: Behavioral: Survey
- Comfort Care Default Arm (Experimental): After receiving a description of an impending delivery of a 23 week gestational infant, participants in this arm were presented with the following information:
  The doctor goes on to say that at this hospital infants born at 23 weeks will receive comfort care, unless their parents object. If you decline comfort care please check the box below:
  Please check if you decline comfort care []
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — Participants were randomized to one of two survey groups. In one arm (resuscitation default arm), resuscitation was presented as the course of action that would be followed unless the participant objected. In the other arm (comfort care default arm), comfort care was presented as the course of action that would be followed unless the participant objected.

SUMMARY:
The purpose of this study is to study how people make decisions regarding delivery room management for infants born extremely premature when survival and long term outcomes are uncertain. The hypothesis is that the way in which information is presented will impact decisions.

There have been many advances in neonatal care in recent decades. However, the investigators do not know if these children will grow up to be healthy or if they will have problems with mental retardation, behavior or physical handicaps. In these circumstances, where the medical profession cannot predict what sort of life a child will have, parents have a choice of having intensive care started or of allowing the baby to die naturally. The age most often cited by physicians at which this care is optional and under parental discretion is 23 weeks gestation.

The purpose of this study was to ask people, recruited through the world wide web, what they would want for the doctor to do in the case of a hypothetical 23 week premature delivery in order to evaluate the decision process and the presence of autonomous choice. This study had two parts. The first part, presented outcome information in 2 different ways -either as survival and lack of severe disability or as mortality and presence of severe disability. The results of the first part have been published (Message Framing and Perinatal Decisions, Pediatrics, 2008). The second part, investigated whether the way in which the way in which delivery room management options were presented- either as agreeing with a course of action or opting out- impacted resuscitation decisions. This part was administered as a separate survey to a different sample of participants at a later date. The remainder of the questionnaires asked demographic and opinion questions as a means to assess variables that may influence how people respond to the information they receive.

ELIGIBILITY:
Inclusion Criteria:

>18 yo

Exclusion Criteria:

<18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2006-05; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Number of participants deciding to resuscitate an extremely premature infant. | Up to 1 year from the start of the study
  Each participants decisional outcome (resuscitation or comfort care) per survey arm will be counted. We expect 60% of the participants will decide to resuscite in both arms. We expect that 90% will select resuscitation in those who receive the resuscitation default and 60% will select resuscitation in the comfort care default

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Murphy, PhD, Principal Investigator — Columbia University; Elke U Weber, Principal Investigator — Columbia University
Locations (1):
- Columbia University Center for Decision Sciences, New York, New York, United States

REFERENCES:
- [Result] Haward MF, Murphy RO, Lorenz JM. Message framing and perinatal decisions. Pediatrics. 2008 Jul;122(1):109-18. doi: 10.1542/peds.2007-0620. PMID 18595993